CLINICAL TRIAL: NCT01748318
Title: New Mexico Honey Wound Treatment Research Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: R. Stephen Rankin, M.D. (Individual)
Responsible Party: Sponsor-Investigator, R. Stephen Rankin, M.D., Primary Investigator, Rankin, R. Stephen, M.D.
Organization: Rankin, R. Stephen, M.D. (Individual)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IND 115653
Record Dates: First submitted 2012-12-10; First posted 2012-12-12 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Community-acquired Methicillin-resistant Staphylococcus Aureus Infection
Keywords: Community acquired MRSA; New Mexico Honey
MeSH Terms: interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NM Regional Honey (Experimental): 15 ml of NM Honey applied directly to wound
  Interventions: Drug: New Mexico Honey; Drug: Bactrim DS
- Bactrim DS (Active Comparator): Standard of Care Oral Antibiotic
  Interventions: Drug: New Mexico Honey; Drug: Bactrim DS

INTERVENTIONS:
Drug: New Mexico Honey — Apply 15 ml of NM Honey to CA-MRSA Abscess compare to standard antibiotic treatment
  Other Names: Local New Mexico Honey
Drug: Bactrim DS — Bactrim DS
  Other Names: sulfamethoxazle-trimethroprim DS

SUMMARY:
In a time of emerging bacteria that are resistant to antibiotics, honey offers an alternative that has potential to reduce the heavy reliance on pharmaceutical antibiotics. We will be evaluating the effectiveness of a locally produced New Mexico Honey against the standard of care Bactrim antibiotic on Community Acquired MRSA.

DETAILED DESCRIPTION:
Locally grown New Mexico Honey will be utilized on abscess wounds of the trunk and extremities vs routine (Bactrim) antibiotic care to determine if NM Honey is effective treatment for Community Acquired MRSA 6 cm abscesses.

ELIGIBILITY:
Inclusion Criteria:

* Patients 16 years of age or older
* Abscess less than or equal to 6 cm in diameter on the extremity or trunk requiring incision and drainage
* Patient willing to try honey prepared dressing
* Patient able to return to office each day for 7 days for evaluation

Exclusion Criteria:

* Under the age of 16
* Abscess of face, scalp or genitals
* Diagnosed as a diabetic
* Allergic to bee pollen, honey or sulfa antibiotics
* Diagnosed with peripheral vascular disease
* Patient acknowledgement of current drug or alcohol abuse

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-03; Primary Completion 2018-05 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Size of lesion at day 7 | 7 days
  Increase in size will determine failure; Decrease in size will determine success

CONTACTS AND LOCATIONS:
Overall Officials: R Stephen Rankin, MD, Principal Investigator
Locations (1):
- Pinon Family Practice, Farmington, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Yes